CLINICAL TRIAL: NCT06300424
Title: Neoadjuvant Almonertinib Followed by Adebrelimab-based Chemo-immunotherapy in II-IIIB EGFR-mutant Non-small Cell Lung Cancer, a Single Arm, Phase II Study
Brief Title: Neoadjuvant Almonertinib Followed by Chemo-immunotherapy in II-IIIB EGFR-mutant NSCLC
Acronym: NEOVADE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-zhao ZHONG, Principal Investigator, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-162
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Non Small Cell Lung Cancer; EGFR Gene Mutation
Keywords: non small cell lung cancer; neoadjuvant therapy; immunotherapy; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; Carboplatin; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Almonertinib and Chemo-immunotherapy (Experimental): 6 weeks of almonertinib followed by 3 cycles of neoadjuvant adebrelimab (1200mg every 3 weeks) with nab-paclitaxel and carboplatin (nab-paclitaxel 135 mg/m2, d1 and d8, and carboplatin AUC 5, d1 every 3 weeks) will be administered before surgery, followed by optional adjuvant treatment including EGFR-TKIs up to 3 years or immunotherapy for up to 1 year or till disease progression or unacceptable toxicity.
  Interventions: Drug: almonertinib; Drug: Carboplatin; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: almonertinib — 110mg qd
Drug: Carboplatin — AUC 5, d1 every 3 weeks
Drug: Nab paclitaxel — 135 mg/m2, d1,d8 every 3 weeks

SUMMARY:
Phase II, single-arm, open-label study that assess clinical feasibility and safety of neoadjuvant almonertinib followed by 3 cycles neoadjuvant adebrelimab plus chemotherapy in EGFR-mutant stage IIA-IIIB NSCLC followed by surgery, adjuvant treatment was upon investigators' decisions.

DETAILED DESCRIPTION:
This study plans to include 32 eligible II-IIIB non small cell lung cancer (NSCLC), patients will receive 6 weeks of almonertinib, and to avoid overlap of interstitial lung disease (ILD) and immune-related pneumonitis, 2 weeks of washout period was designed before 3 cycles of adebrelimab + doublet platinum-based chemotherapy is administered. Dynamic blood samples before, during or after neoadjuvant treatment will be obtained for exploratory analysis. Patients with local disease and resectable or potentially resectable NSCLC will receive anatomic resection. Patients who progress upon neoadjuvant treatment and further assessed as unresectable disease will be scheduled for local radiation or other potential subsequent treatment regarding multidisciplinary discussion. After completion of local treatment (surgery or radiation), patients will undergo optional adjuvant treatment including epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI) or immunotherapy upon investigators' consideration or CT surveillance. Patients will be follow-up within 5 years after surgery. The primary endpoint of this study is major pathological response (MPR) defined as no more than 10% residual tumor found in primary lung cancer as per International Association for the Study of Lung Cancer (IASLC) criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female，Age: 18 Years and older,
2. Subjects voluntarily joined the study and signed informed consent,
3. pathological proven resectable stage II-IIIB non small cell lung cancer (AJCC 8th edition),
4. ECOG PS=0 or 1,
5. resectable or potentially resectable, or resectability discussed by MDT,
6. harboring EGFR mutation: Ex19del, L858R, T790M, G719X, Exon20 insertions, S768I or L861Q
7. measurable lesion as per RECIST1.1.

Exclusion Criteria:

1. pathologica or cytological proven small cell lung cancer, mixed small cell lung cancer or other than non small cell lung cancer,
2. non small cell lung cancer harboring other driver gene alteration with approved targeted drugs,
3. with malignant plural effusion,
4. previous treatment to non small cell lung cancer other than this regimen,
5. received thoracic radiotherapy,
6. currently enrolled in other clinical trial,
7. active or known or suspected autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | MPR will be assessed within 2 weeks after surgery
  MPR was defined as percentage of tumor cells within tumor bed less than 10% for primary lung lesions

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) | pCR will be assessed within 2 weeks after surgery
  The pathological complete response is defined as the absence of residual tumor in both lung and lymph nodes after neoadjuvant treatment.
Objective Response Rate (ORR) | Tumor response will be evaluated within 2 weeks after almonertinib, and within 3-4 weeks after last dose of neoadjuvant treatment
  ORR is the number of participants with a Complete Response (CR) and Partial Response (PR) divided by the total number of participants. Response is based on the Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria. Complete Response (CR) was defined as the disappearance of all target lesions. Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions compared to baseline or the complete disappearance of target lesions, with persistence of 1 or more nontarget lesion(s) and no new lesions.

OTHER OUTCOMES:
Overall Survival (OS) | up to 60 months.
  From date of initiation of neoadjuvant treatment till the date of all-cause death, assessed up to 60 months.
Event Free Survival (EFS) | From date of initiation of neoadjuvant treatment till the date of first documented disease progression or death, whichever came first, assessed up to 60 months
  Time from initiation of neoadjuvant treatment to any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause.
Incidence of Adverse Events (AEs) | up to 90 days.
  Incidence of all grade AE which has been confirmed to be correlated with neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wen-zhao Zhong, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No